CLINICAL TRIAL: NCT06574945
Title: Efficacy and Safety of Propofol in Combination With Different Esketamine Doses for Anesthesia During Loop Electrosurgical Excision Procedure
Brief Title: Anesthesia for Loop Electrosurgical Excision Procedure (LEEP).
Acronym: ESK，LEEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qian Wu (Other)
Responsible Party: Sponsor-Investigator, Qian Wu, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-71
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Esketamine; Loop Electrosurgical Excision; Propofol

STUDY DESIGN:
Intervention Model Description: Patients were categorized into three groups: propofol (2 mg/kg) + normal saline (group P), propofol (1.5 mg/kg) + ESK (0.5 mg/kg) (group PK1), and propofol (1.5 mg/kg) + ESK (0.25 mg/kg) (group PK2). In group P, patients received an intravenous injection of an equivalent dose of normal saline followed by 2 mg/kg of propofol. Group PK1 received an intravenous injection of 0.5 mg/kg ESK followed by 1.5 mg/kg of propofol. Similarly, group PK2 received an intravenous injection of 0.25 mg/kg ESK followed by 1.5 mg/kg of propofol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group P (Placebo Comparator): Intravenous injection of an equivalent dose of normal saline followed by 2 mg/kg of propofol
  Interventions: Drug: intravenous injection of propofol only
- group PK1 (Experimental): Intravenous injection of 0.5 mg/kg esketamine followed by 1.5 mg/kg of propofol
  Interventions: Drug: intravenous injection of propofol +esketamine
- group PK2 (Experimental): Intravenous injection of 0.25 mg/kg esketamine followed by 1.5 mg/kg of propofol
  Interventions: Drug: intravenous injection of propofol +esketamine

INTERVENTIONS:
Drug: intravenous injection of propofol only — Propofol was administered intravenously 2 mg/kg
  Arms: group P
Drug: intravenous injection of propofol +esketamine — intravenous injection of 0.5 mg/kg ESK followed by 1.5 mg/kg of propofol or intravenous injection of 0.25 mg/kg ESK followed by 1.5 mg/kg of propofol
  Arms: group PK1; group PK2

SUMMARY:
The goal of this prospective, randomized controlled study study is to investigate the efficacy and safety of propofol combined with different doses of esketamine (ESK) for anesthesia during loop electrosurgical excision procedure (LEEP).Ninety female patients undergoing LEEP were randomly allocated to three groups.It aims to answer :1.The effect of esketamine combined with propofol in respiration, circulation, etc,during LEEP. 2.The appropriate dosage of esketamine when combined with propofol in LEEP anesthesia.

DETAILED DESCRIPTION:
To investigate the efficacy and safety of propofol combined with different doses of esketamine (ESK) for anesthesia during loop electrosurgical excision procedure (LEEP). Ninety female patients undergoing LEEP were randomly allocated to three groups: group P (2 mg/kg propofol + saline), group propofol + esketamine(PK)1 (1.5 mg/kg propofol + 0.5 mg/kg ESK), and group PK2 (1.5 mg/kg propofol + 0.25 mg/kg ESK). Parameters including mean arterial pressure (MAP), heart rate (HR), respiratory rate (RR), oxygen saturation (SPO2), and venous carbon dioxide (PvCO2) were recorded. Additionally, the need for supplemental propofol, jaw thrust maneuver or ventilation, postoperative awakening time, and adverse reactions were assessed.

ELIGIBILITY:
Inclusion Criteria：

* Patients who will undergo Loop Electrosurgical Excision Procedure
* The age of the patients ranged from 20 to 60 years old
* Paients had a BMI of 18-30 kg/m2
* ASA physical status grade of I or II

Exclusion Criteria:

* Patients who refused to participate
* History of hypertension, hyperthyroidism, or neurological or mental disorder
* Currently taking or has taken opioids and non-steroidal anti-inflammatory drugs within 48 h before surgery
* Participated in other drug clinical trials within 4 weeks
* Allergy to esketamine or propofol
* History of opioid or esketamine addiction

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cervical lesions
Enrollment: 90 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | Immediately upon entering the operating room , 1 and 5 minutes after injection of anesthetics
  The respiratory rate (RR) was monitored from 3-lead ECG
Heart Rate | Immediately upon entering the operating room , 1 and 5 minutes after injection of anesthetics
  The heart rate (HR) was monitored using 3-lead ECG
Mean Arterial Pressure | Immediately upon entering the operating room, 1 and 5 minutes after injection of anesthetics
  The mean arterial pressure (MAP) was monitored using Noninvasive blood pressure monitor
Venous Carbon Dioxide | Immediately upon entering the operating room and 5 minutes after injection of anesthetics
  The venous carbon dioxide (PvCO2) was monitored using blood-gas analyzer

SECONDARY OUTCOMES:
number of additional propofol usage | On the day of surgery, from the instant the anesthesia induction is completed to the instant completion of surgery,up to 10 minutes
  The number of additional propofol was recorded
postoperative awakening time | On the day of surgery, from the instant completion of surgery to the moment the patient wakes up (when MOAA score >4),up to 10 minutes
  The postoperative awakening time (MOAA/S score >4) was recorded
number of jaw thrust maneuver or face mask ventilation | On the day of surgery, from the instant the anesthesia induction is completed to the instant completion of surgery,up to 10 minutes
  The number of jaw thrust maneuver or face mask ventilation was recorded
incidences of postoperative vertigo, nausea, agitation and delirium | On the day of surgery,from the moment the patient wakes up (when MOAA score >4) to the moment the patient leaving the recovery room,up to 30minutes
  incidences of postoperative vertigo, nausea, agitation and delirium were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Gang Y Hao, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan T, Zhang GH, Wang BN, Sun L, Zheng H. Effects of propofol/remifentanil-based total intravenous anesthesia versus sevoflurane-based inhalational anesthesia on the release of VEGF-C and TGF-beta and prognosis after breast cancer surgery: a prospective, randomized and controlled study. BMC Anesthesiol. 2018 Sep 22;18(1):131. doi: 10.1186/s12871-018-0588-3. PMID 30243294
- [Background] Song N, Yang Y, Zheng Z, Shi WC, Tan AP, Shan XS, Liu H, Meng L, Peng K, Ji FH. Effect of Esketamine Added to Propofol Sedation on Desaturation and Hypotension in Bidirectional Endoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2347886. doi: 10.1001/jamanetworkopen.2023.47886. PMID 38117498
- [Background] Oh C, Kim Y, Eom H, Youn S, Lee S, Ko YB, Yoo HJ, Chung W, Lim C, Hong B. Procedural Sedation Using a Propofol-Ketamine Combination (Ketofol) vs. Propofol Alone in the Loop Electrosurgical Excision Procedure (LEEP): A Randomized Controlled Trial. J Clin Med. 2019 Jun 28;8(7):943. doi: 10.3390/jcm8070943. PMID 31261820
- [Background] Eberl S, Koers L, van Hooft J, de Jong E, Hermanides J, Hollmann MW, Preckel B. The effectiveness of a low-dose esketamine versus an alfentanil adjunct to propofol sedation during endoscopic retrograde cholangiopancreatography: A randomised controlled multicentre trial. Eur J Anaesthesiol. 2020 May;37(5):394-401. doi: 10.1097/EJA.0000000000001134. PMID 31860599
- [Background] Jonkman K, van Rijnsoever E, Olofsen E, Aarts L, Sarton E, van Velzen M, Niesters M, Dahan A. Esketamine counters opioid-induced respiratory depression. Br J Anaesth. 2018 May;120(5):1117-1127. doi: 10.1016/j.bja.2018.02.021. Epub 2018 Mar 26. PMID 29661389
- [Background] Nie J, Chen W, Jia Y, Zhang Y, Wang H. Comparison of remifentanil and esketamine in combination with propofol for patient sedation during fiberoptic bronchoscopy. BMC Pulm Med. 2023 Jul 11;23(1):254. doi: 10.1186/s12890-023-02517-1. PMID 37430293
- [Background] Trujillo KA, Heller CY. Ketamine sensitization: Influence of dose, environment, social isolation and treatment interval. Behav Brain Res. 2020 Jan 27;378:112271. doi: 10.1016/j.bbr.2019.112271. Epub 2019 Oct 5. PMID 31593791

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT06574945/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT06574945/ICF_001.pdf